CLINICAL TRIAL: NCT05125107
Title: PrOgnostic imPlicaTIons of 2-diMensIonal Patterns for Residual Disease After Stenting CharacteriZEd by Quantitative Flow Ratio Pullback Curve Analysis
Acronym: CHART-OPTIMIZE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-20211112
Record Dates: First submitted 2021-11-17; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Predominant focal residual disease without major gradient
  Interventions: Device: Quantitative Flow Ratio derived PPG and dQFR/ds
- Group 2: Predominant focal residual disease with major gradient
  Interventions: Device: Quantitative Flow Ratio derived PPG and dQFR/ds
- Group 3: Predominant diffuse residual disease without major gradient
  Interventions: Device: Quantitative Flow Ratio derived PPG and dQFR/ds
- Group 4: Predominant diffuse residual disease with major gradient
  Interventions: Device: Quantitative Flow Ratio derived PPG and dQFR/ds

INTERVENTIONS:
Device: Quantitative Flow Ratio derived PPG and dQFR/ds — From coronary angiographic images, QFR will be calculated and virtual pullback curve will be abstracted and PPG index will be calculated as:
  PPG index={MaxPPG20mm/△QFRvessel+(1-length with functional disease/Total vessel length) }/2
  Physiologic local severity of coronary atherosclerosis was assessed by instantaneous QFR gradient per unit length (dQFR/ds)

SUMMARY:
The purpose of this study is to investigate the prognostic values of 2-dimensional residual disease patterns determined by quantitative flow ratio (QFR) pullbacks after stent implantation.

DETAILED DESCRIPTION:
Prognostic value of post-percutaneous coronary intervention (PCI) percutaneous coronary intervention (PCI) physiology assessment has been confirmed. The rationale for measuring post-PCI physiologic outcome is that it could implicate the residual risk of suboptimal stenting in addition to residual diffuse coronary artery disease after PCI Nevertheless, it should be noted that both post-PCI physiologic indices such as ,fractional flow reserve (FFR) and QFR, are measured at the distal of the interrogated vessel and reflect the cumulative residual disease burdens, defining the residual disease patterns might have additional role in exploring the underlying mechanisms for suboptimal post-PCI physiologic results, thus providing the opportunities for functional optimization with subsequent interventions accordingly to improve immediate functional results, long-term outcomes may be positively affected.

Concept of physiologic 2-dimensional disease patterns according to both physiologic distribution (predominant focal versus diffuse disease) and local severity (presence versus absence of major gradient) of coronary atherosclerosis before PCI was proposed and could be derived from virtual QFR pullback curve. Nevertheless, the prognostic value of the 2-dimensional residual disease patterns after PCI has not been studied yet.

The CHART-OPTIMIZE study aims to investigate the clinical implications of physiologic 2-dimensional residual disease patterns after stenting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one vessel with measurable post-PCI QFR
* PPG index can be calculated from virtual QFR pullback curve
* dQFR/ds can be calculated from virtual QFR pullback curve
* The patient is willing to comply with specified follow-up evaluations;
* Patients who agree to accept the follow-up visits.

Exclusion Criteria:

* Culprit vessels for ACS myocardial infarction;
* Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following index procedure;
* Patient has other medical illness (e.g., cancer, known malignancy, congestive heart failure, organ transplant recipient or candidate) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e., less than 1 year);
* Patient has a known hypersensitivity or contraindication to aspirin, heparin, clopidogrel/ticlopidine, stainless steel alloy, cobalt chromium, rapamycin, styrene-butylenes-styrene or poly-lactic acid (PLA) polymer, and/or contrast sensitivity that cannot be adequately pre-medicated;
* Any significant medical condition which in the Investigator's opinion may interfere with the patient's optimal participation in the study;
* Currently participating in another investigational drug or device study or patient in inclusion in another investigational drug or device study during follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All vessels with measurable post-PCI QFR and with available post-PCI QFR virtual pullback curves were included
Sampling Method: Non-Probability Sample
Enrollment: 1607 (Estimated)
Dates: Start 2021-11-15 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Vessel-oriented composite outcome | at 2 years from index procedure
  Vessel-oriented composite outcome (VOCO) including vessel related ischemia-driven target vessel revascularization, vessel-related myocardial infarction (MI), and cardiac death.

SECONDARY OUTCOMES:
Cardiac death or vessel-related MI | at 2 years from index procedure
  Cardiac death or vessel-related MI
Vessel-related MI | at 2 years from index procedure
  Vessel-related MI
Cardiac death | at 2 years from index procedure
  Cardiac death
Ischemia-driven target vessel revascularization | at 2 years from index procedure
  Ischemia-driven target vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Professor, Study Chair — Fudan University; Bo Xu, MBBS, Principal Investigator — Fu Wai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu B, Gao R, Yang Y, Cao X, Qin L, Li Y, Li Z, Li X, Lin H, Guo Y, Ma Y, Wang J, Nie S, Xu L, Cao E, Guan C, Stone GW; PANDA III Investigators. Biodegradable Polymer-Based Sirolimus-Eluting Stents With Differing Elution and Absorption Kinetics: The PANDA III Trial. J Am Coll Cardiol. 2016 May 17;67(19):2249-2258. doi: 10.1016/j.jacc.2016.03.475. PMID 27173037
- [Background] Dai N, Hwang D, Lee JM, Zhang J, Jeon KH, Paeng JC, Cheon GJ, Koo BK, Ge J. Feasibility of Quantitative Flow Ratio-Derived Pullback Pressure Gradient Index and Its Impact on Diagnostic Performance. JACC Cardiovasc Interv. 2021 Feb 8;14(3):353-355. doi: 10.1016/j.jcin.2020.10.036. No abstract available. PMID 33541549
- [Background] Dai N, Zhang R, Hu N, Guan C, Zou T, Qiao Z, Zhang M, Duan S, Xie L, Dou K, Zhang Y, Xu B, Ge J. Integrated coronary disease burden and patterns to discriminate vessels benefiting from percutaneous coronary intervention. Catheter Cardiovasc Interv. 2022 Jan 1;99(1):E12-E21. doi: 10.1002/ccd.29983. Epub 2021 Oct 15. PMID 34652068